CLINICAL TRIAL: NCT05273021
Title: Implementation and Validation of the Dutch Translation of the TAPS-tool: a Screener for Tobacco, Alcohol, Prescription Medication and Other Substances for Patients With Severe Mental Illness With and Without Intellectual Disability
Brief Title: Validation of the Dutch Translation of the Tobacco, Alcohol, Prescription Medication and Other Substances (TAPS)-Tool
Status: Recruiting | Type: Observational
Sponsor: Birgit Seelen-de Lang (Other)
Collaborators: Ggz Oost Brabant (Other)
Responsible Party: Sponsor-Investigator, Birgit Seelen-de Lang, Psychologist, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Other Study IDs: ECSW-2021-051
Record Dates: First submitted 2022-02-11; First posted 2022-03-10 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Substance Use; Severe Mental Disorder; Intellectual Disability, Mild
Keywords: TAPS; screener
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders; Intellectual Disability; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- participants with substance use problems: There are 2 subgroups:
  * Participants without intellectual disabilities
  * Participants with intellectual disabilities with and without severe mental illness
  Interventions: Diagnostic Test: TAPS

INTERVENTIONS:
Diagnostic Test: TAPS — all participants are investigated by the Dutch TAPS tool (Tobacco, Alcohol, Prescription medication and other Substances-tool). A screener and short assessment of possible substance use problems

SUMMARY:
The aim of the study is to investigate the reliability and validity of the Dutch version of the TAPS-tool.

This will be investigated in 2 groups: patients without intellectual disabilities treated in Flexible Assertive Community Treatment (FACT) teams and patients with intellectual disabilities. For the later group, an adjusted version of the TAPS-tool will be developed.

For both groups the TAPS outcome will be compared to a golden standard.

DETAILED DESCRIPTION:
All FACT teams in the participating organization (GGZ Oost Brabant) work through a standardized care pattern which implicates screening and assessment on several areas. At the start of the treatment all patients are assessed for intellectual disabilities, trauma related symptoms, addiction, quality of life, level of psychiatric complaints, social functioning, and phase of recovery. Subsequently quality of life and the level of psychiatric complaints is measured yearly. For this research question a small golden standard instrument was added to the standard screening and assessment.

For people with intellectual disabilities (ID) who get an extensive assessment of substance use problems in their (standard) treatment, permission to participate on the TAPS (version for ID) was asked.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated in the participating FACT teams and for patients treated at the LVB-P (department for patients with intellectual disabilities and psychiatric disorders [Dutch name]) department of the GGZ Oost Brabant or the ORO foundation (ORO is no abbreviation but just a name of the institute).

Exclusion Criteria:

* If patients do not have sufficient command of the Dutch language or cannot concentrate for 20 minutes, the instruments are not taken

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: secondary psychiatric care departments and special services for people with intellectual disabilities
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
TAPS | one assessment at the start of the treatment
  The TAPS-tool is a 2-phase screening instrument to detect substance use problems which can be used as an interview or as a self-administered questionnaire. TAPS 1 has a score from 0-4 (higher is more substance use). For a score of 1 or higher, TAPS 2 is also taken. TAPS 2 has a total score from 0-3 (higher is indication of more problematic use) for all of the 8 substances. Cut off score is +2.
Measurement of Addiction for Triage and Evaluation (MATE) | At the start of FACT treatment, only for participants of this study
  MATE is an instrument, developed in Europe to determine patient characteristics for the indication of care for people with addiction problems on a valid and reliable way. The MATE will be used for participants without intellectual disabilities. Modules 1, 4, and Q1 are used in this study.
  Module 1 (interview about substance use) for alcohol, nicotine, cannabis, opiates, cocaine, stimulant drugs, extacy, other drugs, sedative medicines and gambling. For every substance there is a cut off point for excessive use. There are no scores for module 1.
  Module 4: 11 binary questions (yes/no) about dependency and misuse of the problem area. The scoring range is 0 to 9 (cut off = 8). the higher the score, the worse the dependency.
  Module Q1: five questions about desire, based on a five point Likert-scale (score 0-4). Cut off = sum score > 12. higher scores stand for more problematic desire.
Substance use measurement for people with intellectual disabilities (SumID-Q) | Standard assessment at the start of the treatment, or when substance use problems are suspected
  The SumID-Q is an extensive Dutch assessment instrument (interview) on substance use problems for people with intellectual disabilities. There are no total scores.

SECONDARY OUTCOMES:
Health of the Nation Outcome Scales (HoNOS) | Once at start of FACT treatment
  The Health of the Nation Outcome Scales (HONOS] is a scaling device routinely used by the mental health services in Anglo-Saxon countries in order to map a patient's mental state and any changes that may have occurred in it. The 12 questions are scored from 0-4. 0 = no problems; 4 = very serious problems. Psychometric properties of the HoNOS are satisfactory to good (Mulder et al., 2004). There is a total sum score available (and reference group: patients with severe mental illness)..
Manchester abbreviated quality of life measure (MANSA) | Once, at start of FACT treatment
  Self administered questionnaire on quality of life. The MANSA is a multi-dimensional questionnaire which consists of 16 items. Twelve items determine patient satisfaction with their life as a whole, employment, financial situation, number and quality of friendships, leisure activities, accommodation, personal safety, social network, sex life, relationship with family, physical health and mental health. Satisfaction on these items is rated on a seven-point rating scale (1 = extremely negative, 7 = extremely positive). Four objective items assess the existence of a 'close friend', whether there was contact with a friend in the last week, accusation of a crime, and victimization of physical violence (yes / no). These objective items do not count in the calculation of the total score. In this research, the summed scores were used.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - GGZ Oost Brabant - FACT, Boekel, North Brabant
  - GGZ Oost Brabant - LVB-P, Boekel, North Brabant
  - Stichting ORO, Helmond, North Brabant

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT05273021/Prot_SAP_000.pdf
  • Informed Consent Form: ICF FACT (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT05273021/ICF_001.pdf
  • Informed Consent Form: ICF LVB-P (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT05273021/ICF_002.pdf
  • Informed Consent Form: ICF ORO (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT05273021/ICF_003.pdf